CLINICAL TRIAL: NCT03997643
Title: Preservation of Swallowing in Resected Oral Cavity Squamous Cell Carcinoma: Examining Radiation Volume Effects: A Randomized Trial
Brief Title: Preservation of Swallowing in Respected Oral Cavity Squamous Cell Carcinoma: Examining Radiation Volume Effects (PRESERVE): A Randomized Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRESERVE
Record Dates: First submitted 2019-06-14; First posted 2019-06-25 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Head and Neck Cancer
Keywords: Radiation Therapy; Oral Cavity Squamous Cell Carcinoma; Randomized Trial
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Radiotherapy (Active Comparator): Radiotherapy to all dissected areas
  Interventions: Radiation: Radiotherapy to all dissected areas
- Radiotherapy to smaller treatment area (Experimental): Omit radiation to pN0 neck
  Interventions: Radiation: Omit radiation to pN0 neck

INTERVENTIONS:
Radiation: Radiotherapy to all dissected areas — Post operative radiation therapy +/- chemotherapy based on historic treatment volumes (including the primary site, dissected areas +/- elective areas
  Arms: Standard Radiotherapy
Radiation: Omit radiation to pN0 neck — post operation radiation therapy +/- chemotherapy that avoids targeting the dissected pN0 neck
  Arms: Radiotherapy to smaller treatment area

SUMMARY:
The goal of this randomized treatment study is to formally compare quality of life in patients with at least one pN0 hemi-neck after resection of a squamous cell carcinoma of the oral cavity treated with a primary radiation therapy versus a secondary targeted radiation therapy approach, to provide a high level of evidence to guide the selection of treatment options.

DETAILED DESCRIPTION:
The goal of this randomized treatment study is to formally compare quality of life in patients with at least one pN0 hemi-neck after resection of a squamous cell carcinoma of the oral cavity treated with a primary radiation therapy versus a secondary targeted radiation therapy approach, to provide a high level of evidence to guide the selection of treatment options.

The study will require a sample size of 90 patients randomized in a 2:3 between the two arms. Arm 1 (standard radiation therapy to tumor location and surrounding area) and Arm 2 (targeted radiation therapy to tumor location).

Patients will be followed for a total of 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Willing to provide informed consent
* ECOG performance status 0-2
* Histologically confirmed, resected oral cavity squamous cell carcinoma with at least ipsilateral selective neck disection
* Patient has pathological features that are indications for PORT: positive or close (≤ 3 mm) margin, presence of LVI or PNU, pT3 or pT4 disease, positive lymph nodes, and PORT is recommended by treating physician
* Pathologically lympth node negative in at least one dissected hemi-neck with at least 10 nodes recovered in each pN0 hemi-neck

Exclusion Criteria:

* Serious medical comorbidities or other contraindications to radiotherapy
* Prior history of head and neck cancer within 5 years
* Any other active invasive malignancy, except non-melanotic skin cancers
* Prior head and neck radiation at any time
* Prior oncologic head and neck surgery in the oral cavity or neck
* Metastatic disease
* Locoregional disease recurrence identified following surgical resection but prior to the start of radiotherapy
* Inability to attend full course of radio therapy or follow-up visits
* Unable or unwilling to complete QoL questionnaires
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-09-06 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Regional failure in the pN0 hemi-neck (s) | Baseline to 5 years
  Rate of relapse in the pN0 neck in Arm 2 compared to historical controls

SECONDARY OUTCOMES:
Swallowing Quality of life | Baseline up to 12 months
  Assessed with the MD Anderson Dysphagia Inventory (MDADI) scale
Swallowing Quality of life | Baseline up to 12 months
  Assessed with the EORTC QLQ-C30 scale
Swallowing Quality of life | Baseline up to 12 months
  Assessed with the EORTC QLQ H&N 35 scale
Health Status Quality of life | Baseline up to 12 months
  Assessed with the EORTC EQ-5D-5L scale
Overall survival | Baseline to 5 years
  Defined as time from randomization to death from any cause
Disease free survival | Baseline to 5 years
  Defined as the measure of time after treatment during which no sign of cancer is found
Local recurrence | Baseline to 5 years
  Defined as Cancer that has recurred at or near the same place as the primary tumor, usually after a period of time during which the cancer could not be detected.
Regional recurrence | Baseline to 5 years
  Defined as recurrence that occurs in the lymph nodes and tissue located in the vicinity of your original cancer
Locoregional recurrence | Baseline to 5 years
  Defined as the recurrence of cancer cells at the same site as the original tumor and/or the regional lymph nodes after a disease free period.
Rate of salvage treatment (surgery +/- radiotherapy) in the pN0 neck and freedom from unsalvageable neck recurrence | Baseline 5 years
  Rate of salvage treatment (surgery +/- radiotherapy) in the pN0 neck and freedom from
Rate of feeding tub insertion and rate of feeding tube use at 1-year post randomization | Randomization to 1 year post randomization
  Rate of feeding tub insertion and rate of feeding tube use at 1-year post randomization
Swallowing function | Baseline to 1 year
  Measured by the Modified Barium Swallow Impairment (MBsimp) score
Swallowing function | Baseline to 1 year
  Measured by the Dynamic Imaging Grade of Swallowing Toxicity score
Swallowing function | Baseline to 1 year
  Measured by the Functional Oral Intake Score
Rate of toxicity | Baseline to 5 years
  Assessed using the National Cancer Institute Common Toxicity Criteria (NCI-CTC) version 4
Rate of failure in the clinically node negative neck | Baseline to 5 years
  defined as time from randomization to failure in the cN0 neck

CONTACTS AND LOCATIONS:
Locations (8):
- Miami Cancer Institute, Miami, Florida, United States
- Canada (2):
  - London Regional Cancer Program, London, Ontario
  - CHUM, Montreal, Quebec
- Ireland (4):
  - Cork University Hospital, Wilton, County Cork
  - University Hospital Galway, Newcastle Road, Galway, County Galway
  - St. Luke's Radiation Oncology Network, Rathgar, Dublin
  - Beaumont St. Luke's Centre, Dublin, Leinster
- Beatson West of Scotland Cancer Centre, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lang P, Contreras J, Kalman N, Paterson C, Bahig H, Billfalk-Kelly A, Brennan S, Rock K, Read N, Venkatesan V, Sathya J, Mendez LC, MacNeil SD, Nichols AC, Fung K, Mendez A, Winquist E, Kuruvilla S, Stewart P, Warner A, Mitchell S, Theurer JA, Palma DA. Preservation of swallowing in resected oral cavity squamous cell carcinoma: examining radiation volume effects (PRESERVE): study protocol for a randomized phase II trial. Radiat Oncol. 2020 Aug 14;15(1):196. doi: 10.1186/s13014-020-01636-x. PMID 32795322